CLINICAL TRIAL: NCT02434614
Title: A Randomized Phase III Non-inferiority Study of Induction Chemotherapy Followed by IMRT Alone Versus Induction Chemotherapy Followed by IMRT Plus Concurrent Chemotherapy in Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Induction Chemotherapy Followed by IMRT With or Without Concurrent Chemotherapy in Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wei Jiang (Other)
Collaborators: Wuzhou Red Cross Hospital (Other); Guangxi Naxishan Hospital (Other); LiuZhou People's Hospital (Other); Guigang People's Hospital (Other); Youjiang Medical College for Nationalities (Other); Nanning Monority Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Wei Jiang, Ph.D., Guilin Medical University, China
Organization: Guilin Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLMU-01
Record Dates: First submitted 2015-04-27; First posted 2015-05-05 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Docetaxel; CF regimen; Radiotherapy, Intensity-Modulated; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Induction CT+IMRT alone (Experimental): Induction Chemotherapy(CT) Followed by Intensity-modulated Radiation Therapy (IMRT )alone
  Interventions: Drug: Docetaxel,Cisplatin,Fluorouracil; Radiation: Intensity-modulated radiation therapy (IMRT)
- Induction CT+IMRT Combined Concurrent CT (Active Comparator): Induction Chemotherapy(CT) Followed by Intensity-modulated Radiation Therapy (IMRT ) Combined Concurrent Chemotherapy
  Interventions: Drug: Docetaxel,Cisplatin,Fluorouracil; Radiation: Intensity-modulated radiation therapy (IMRT); Drug: Cisplatin

INTERVENTIONS:
Drug: Docetaxel,Cisplatin,Fluorouracil — Induction chemotherapy: patients receive 60 mg/m2 docetaxel intravenously on day 1, 60 mg/m2 cisplatin intravenously on day 1, and 600 mg/m2/d fluorouracil as a continuous infusion on days 1-5; three cycles were administered at intervals of 3 weeks.
  Other Names: No.
Radiation: Intensity-modulated radiation therapy (IMRT) — IMRT is given as 2.0-2.3 Gy per fraction with five daily fractions per week for 6-7 weeks, Cumulative doses were > 66 Gy to the primary tumor and > 50 Gy to the bilateral cervical lymph nodes and potential sites of local infiltration.
  Other Names: No.
Drug: Cisplatin — Concurrent chemotherapy: patients received weekly intravenous cisplatin at 30 mg/m2 for 6-7 weeks.
  Other Names: No.
  Arms: Induction CT+IMRT Combined Concurrent CT

SUMMARY:
Several prospective randomized trials have demonstrated that concurrent chemoradiotherapy was superior to radiotherapy alone in the treatment of locoregionally advanced nasopharyngeal carcinoma (NPC). Based on these evidences, concurrent chemoradiotherapy (CCRT) with/without sequential chemotherapy has become the standard care for locoregionally advanced NPC. However, most of these evidences of standard treatment for locoregionally advanced NPC were based on the two-dimensional conventional radiotherapy (2DCRT). As the intensity-modulated radiation therapy (IMRT) technique has been widely used in the last decades, IMRT improved the treatment outcomes of patients with NPC, especially the local control rate. Currently, more retrospective studies compared the IMRT alone vs. IMRT plus concurrent chemotherapy, and reported that concurrent chemotherapy failed to improve survival rates for patients with locoregionally advanced disease, but increased the severity of acute toxicities. People started to reconsider the role of CCRT. Therefore, we propose this randomized phase III non-inferiority study to reassess the efficacy and contribution of concurrent chemotherapy in locoregionally advanced NPC during IMRT era.

DETAILED DESCRIPTION:
Patients with with previously untreated non-metastatic newly histologically-confirmed non-keratinizing III-IVb NPC (UICC/AJCC 7th edition) are randomly assigned to receive induction chemotherapy followed by IMRT alone (investigational group) or induction chemotherapy followed by IMRT plus concurrent chemotherapy (control group). During induction chemotherapy, patients in both groups receive 60 mg/m2 docetaxel intravenously on day 1, 60 mg/m2 cisplatin intravenously on day 1, and 600 mg/m2/d fluorouracil as a continuous infusion on days 1-5; three cycles were administered at intervals of 3 weeks. During radiotherapy, patients in investigational group received IMRT alone and patients in control group received IMRT, concurrently with weekly intravenous cisplatin at 30 mg/m2 for 6-7 weeks. IMRT is given as 2.0-2.3 Gy per fraction with five daily fractions per week for 6-7 weeks, Cumulative doses were > 66 Gy to the primary tumor and > 50 Gy to the bilateral cervical lymph nodes and potential sites of local infiltration. The primary endpoint is failure-free survival(FFS). Secondary clinical endpoints include overall survival (OS), locoregional failure-free survival (LRFFS), distant failure-free survival (DFFS) rates and toxic effects.

ELIGIBILITY:
Inclusion Criteria:

Patients with newly histologically confirmed non-keratinizing (according to WHO histologically type); Tumor staged as III-IVb (according to the 7th AJCC edition); No pregnant female; Age between 18-70; Normal complete blood count level (hemoglobin >10 g/dL, white blood cells ≥4000/μL, platelets ≥100 000/μL); Normal hepatic functions (serum total bilirubin ≤1.6 mg/dL, serum transminase < 2.5 times higher than upper limit); Normal renal function (serum creatinine ≤1.5 mg/dL, creatinine clearance ≥60 mL/min); Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; Without radiotherapy or chemotherapy; Patients must give signed informed consent.

Exclusion Criteria:

Disease progression in the process of the treatment; The presence of uncontrolled life-threatening illness; History of previous radiotherapy or chemotherapy; Pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2015-03; Primary Completion 2021-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 3 years
  Progression-free survival is to first disease progression [local recurrence and/or distant metastasis] or death from any cause.

SECONDARY OUTCOMES:
Overall Survival | 3 years
  Overall survival is from randomization to death of any cause or last follow-up.
Locoregional Failure-free Survival | 3 years
  Locoregional failure-free survival is from randomization to locoregional progression.
Distant Failure-free Survival | 3 years
  Distant failure-free survival is from randomization to first distant metastasis.
Number of Participants with Adverse Events | 3 years
  Incidence of acute and late toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, Ph.D., Study Director — Guilin Medical University Affiliated Hospital
Locations (6):
- China (6):
  - Affiliated Hospital of Youjiang Medical University for Nationalities, Baise City, Guangxi
  - Guigang People's Hospital, Guigang, Guangxi
  - Guangxi Naxishan Hospital, Guilin, Guangxi
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Nanning Monority Hospital, Nanning, Guangxi
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi

REFERENCES:
- [Derived] Dai J, Zhang B, Su Y, Pan Y, Ye Z, Cai R, Qin G, Kong X, Mo Y, Zhang R, Liu Z, Xie Y, Ruan X, Jiang W. Induction Chemotherapy Followed by Radiotherapy vs Chemoradiotherapy in Nasopharyngeal Carcinoma: A Randomized Clinical Trial. JAMA Oncol. 2024 Apr 1;10(4):456-463. doi: 10.1001/jamaoncol.2023.6552. PMID 38329737